CLINICAL TRIAL: NCT02010008
Title: Understanding and Preventing Breast Cancer Disparities in Latinas: Screening Mammography and Latinas: A Multilevel Intervention
Brief Title: Screening Mammography and Latinas: A Multilevel Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IR 7124; P50CA148143 (NIH)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; cancer disparities; Latino women; Hispanic women; mammography; multi-level intervention
MeSH Terms: conditions — Breast Neoplasms | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing Intervention (Experimental): Motivational Interviewing (MI) Intervention includes in -person home visit that elicits behavior change by helping participants explore and resolve ambivalence. A telephone follow-up call also uses MI technique.
  Interventions: Behavioral: Motivational Interviewing Intervention
- Comparison (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Motivational Interviewing Intervention — An individual-level intervention that implements a motivational interviewing intervention led by a promotora
  Arms: Motivational Interviewing Intervention

SUMMARY:
¡Fortaleza Latina! is a multi-level randomized trial to increase participation in mammography screening among Latinas who seek care at a community health center in Western Washington.

In partnership with the partnering community health center, we have obtained lists of women patients aged 42 to 74 years old who had not had a mammogram in the last two years and resided within defined radii of the four clinics. Baseline and one year follow-up surveys will be obtained by in person home interview. Participants are randomized within clinic to intervention or comparison group. The intervention consist of two motivational interviewing sessions, one in person in the home, and one telephone follow-up. The study hypothesis is that a higher proportion of participants in the motivational interviewing arm will obtain a screening mammogram within the study period than those in the comparison arm.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among Hispanic women in the United States (US) and five-year survival from breast cancer is lower in Hispanic than in non-Hispanic White women. This reduced survival has a number of potential causes, but differential screening rates may be a partial explanation, since Hispanic women have lower breast cancer screening rates than non-Hispanic White women. The overall purpose of the study is to develop and evaluate a culturally-appropriate intervention aimed at increasing screening mammography rates in a clinic-based sample of predominantly Mexican American women in Western Washington.

The recruitment goal of the Fortaleza Latina study is approximately 500 Latina women aged 40-74 who have had a clinic visit within the past 5 years, but no recent mammogram, from the four selected Community Health Center clinics. After providing informed consent and completing a baseline assessment, eligible women are randomly assigned to intervention or comparison group, within clinic. The individual-level intervention implements motivational interviewing (MI) in two participant encounters. MI is a direct counseling style, led by a promotora (lay health advisor), that elicits behavior change by helping participants explore and resolve ambivalence.

Of the 2194 women contacted by field interviewers, a total of 710 surveys have been completed; of these, 542 were eligible and have been randomized and enrolled into the Fortaleza Latina study (279 intervention, 263 usual care).

ELIGIBILITY:
Inclusion Criteria:

* Hispanic/Latina ethnicity
* Have been seen in one of the 4 community clinics in the past 5 years
* have NOT had a mammogram within the past two years
* Residing within 20 miles of one of the participating clinics

Exclusion Criteria:

* Participants who do not match the Eligibility Criteria listed above
* Medical record verified recent mammogram

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2010-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Mammography Screening | One year post baseline
  Through medical record review at one year follow up, women will be classified as receiving or not receiving mammography screening since baseline assessment

SECONDARY OUTCOMES:
Self-report of mammography screening | One year post baseline
  At the one year follow-up women are asked have they ever had a mammogram, and then when was the most recent mammogram. responses are used in conjunction with date of baseline survey.

OTHER OUTCOMES:
Relative cost | one year
  Cost of intervention is set against potential savings in treatment costs associated with late diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Shirley AA Beresford, PhD, Principal Investigator — Fred Hutchinson Cancer Center; Gloria D Coronado, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Coronado GD, Jimenez R, Martinez-Gutierrez J, McLerran D, Ornelas I, Patrick D, Gutierrez R, Bishop S, Beresford SA. Multi-level Intervention to increase participation in mammography screening: inverted exclamation markFortaleza Latina! study design. Contemp Clin Trials. 2014 Jul;38(2):350-4. doi: 10.1016/j.cct.2014.06.008. Epub 2014 Jun 18. PMID 24952281